CLINICAL TRIAL: NCT02955277
Title: The Effectiveness of TECH: Tablet Enhancement of Cognition and Health, Cognitive Training Using Touchscreen Tablet Gaming Applications, for Older Adults With Mild Cognitive Impairment
Brief Title: The Effectiveness of TECH: Tablet Enhancement of Cognition and Health
Acronym: TECH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Principal Investigator, Zvi Buckman, Dr. Zvi Buckman, Assuta Hospital Systems
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016009-1
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-08

CONDITIONS: Mild Cognitive Impairment
Keywords: Cognitive training; Tablet computers
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors were blind to group allocation.
Oversight: Data Monitoring Committee: No

ARMS (2):
- TECH protocol (Experimental): TECH protocol - Daily self-training using tablet apps facilitated by weekly group sessions. The self-training will take place independently at participants' home and will include mostly playing puzzle-apps to train different cognitive components. Participants will be requested to play (and log) various apps three to five times a week for 30-60 minutes each time, for a total of 15-25 training sessions. In addition they will use the tablets for a variety of everyday uses. The individual self-training will be accompanied by six weekly sessions (of 60 minutes) in a small group setting (5-6 participants) led by an experienced occupational therapist.
  Interventions: Other: TECH: Tablet Enhancement of Cognition and Health protocol
- standard care or active standard care (Active Comparator): Participants will receive standard occupational therapy with no TECH protocol. or Will receive active standard care: six weekly group sessions (60 minutes) for cognitive training using puzzle games. The setting will includes small groups of 5-6 participants, with no self training at home.
  Interventions: Other: Standard care or active standard care

INTERVENTIONS:
Other: TECH: Tablet Enhancement of Cognition and Health protocol — Cognitive training using touchscreen tablets (TECH protocol)
  Arms: TECH protocol
Other: Standard care or active standard care — standard occupational therapy or 6-weekly group sessions playing board games and puzzles.
  Arms: standard care or active standard care

SUMMARY:
This study assess the effectiveness of novel cognitive intervention utilizing tablet apps (TECH protocol: Tablet Enhancement of Cognition and Health) to improve cognitive abilities, daily function and health-related quality of life of older adults with MCI. Older adults with MCI will be randomly allocated to the TECH protocol (experimental group) or standard care (control group). Assessments will be administered pre and post the 6-week TECH protocol and at 6-month follow-up by assessors blind to group allocation.

DETAILED DESCRIPTION:
A single-blind randomized controlled trial (RCT) will be conducted, by assessors blind to group allocation. Participants will be referred to the study from 'Maccabi Healthcare Services' by family physicians and geriatric physician of 'Maccabi Healthcare Services Central District'. The majority of TECH protocol training will take place in the participants' home as self-practice. The assessment and weekly group meetings will take place at clinics of Maccabi Healthcare Services in the Central District. A Helsinki approval (#2016009) has already been obtained. Participants will receive information regarding the study and if eligible will sign a consent form, undergo the screening and then the pre-intervention assessments. Then they will be randomly allocated into experimental or control group by a computer program (stratification of the severity of the cognitive decline according to the Montreal Cognitive Assessment (MoCA) scores of above or below 23 points). The experimental group participants will receive the TECH protocol, while participants in the control group will continue to receive standard care. Following the intervention a second assessment will be performed, as well as six-months follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 and above.
* Have MCI (as determined by the following four criterions: A. a score of 19-25 on the MoCA, B. subjective memory complaints, and report from an informant of the same memory complains (the informant should be a person who interacts with the participant three or more times a week), C. Informant report of the cognitive decline as newly acquired, D. independence in Basic Activities of Daily Living (BADL) and Instrumental Activities of Daily Living (IADL), as reported by the participants and the informant, excluding motor difficulties which are not caused due to neurological conditions or lack of performance with no changes compared to the past.
* Have normal or corrected vision and hearing.
* Speak, write and read Hebrew.
* Able to understand and follow use of the touchscreen of a tablet after initial demonstration.

Exclusion Criteria:

* Experience severe depressive symptoms (10 points or more in The Geriatric Depression Scale)
* Are diagnosed with dementia, or other neurological or psychiatric condition (such as stroke, Parkinson's disease).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zvi Buckman, MD, Principal Investigator — Maccabi Healthcare Services, Israel
Locations (1):
- Maccabi Healthcare Services, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Pre-Post Intervention
Arm/Group | TECH Protocol | Standard Care or Active Standard Care
Started | 30 | 31
Completed | 25 | 25
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 5 | 6
Period: Post to Follow-up
Arm/Group | TECH Protocol | Standard Care or Active Standard Care
Started | 25 | 25
Completed | 17 | 14
Not Completed | 8 | 11
Not completed — Lost to Follow-up | 8 | 11

BASELINE CHARACTERISTICS:
Population: According to the inclusion criteria, all participants had MCI, were independent in BADL and IADL without severe depressive symptoms. Most participants reported to use a smartphone or/and a computer on a daily basis prior to the study, a few reported previous touchscreen tablet experience.
Groups:
- Total: Total of all reporting groups
Arm/Group | TECH Protocol | Standard Care or Active Standard Care | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.6 (5.8) | 75.1 (6.0) | 75.3 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 16 | 17 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Jewish | 30 | 31 | 61
Region of Enrollment [Number; unit: participants]
  Israel | 30 | 31 | 61
Montreal Cognitive Assessment (MoCA) [Mean (Standard Deviation); unit: units on a scale] — This is a cognitive screening tool that assesses global cognition and includes the cognitive components: attention and concentration, executive functions, memory, language, visuo-constructional skills, conceptual thinking, calculations, and orientation.
  scores range from 0-30. A higher score indicates a better cognitive status. A score above 26 indicates normal cognition
  units on a scale | 22.6 (1.8) | 22.3 (1.9) | 22.5 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: The Montreal Cognitive Assessment (MoCA)
Description: A cognitive screening tool that assesses global cognition and includes the cognitive components: attention and concentration, executive functions, memory, language, visuo-constructional skills, conceptual thinking, calculations, and orientation.
  Total score range from 0-30. A higher score indicates a better cognitive status.
  A score above 26 indicates normal cognition
Time Frame: pre intervention, post 5 weeks intervention, follow-up after 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TECH Protocol | Standard Care or Active Standard Care
Number analyzed (Participants) | 30 | 31
units on a scale
  Pre intervention | 22.6 (1.8) | 22.3 (1.9)
  Post 5 week intervention | 23.1 (2.7) | 21.9 (2.5)
  Follow-up after 6 months | 23.3 (3.2) | 21.5 (2.7)

2. Secondary Outcome: WebNeuro
Description: A computerized web-based battery assessment of neurocognitive functioning. The battery will include seven subtests that examine three cognitive domains: memory (Memory recognition/verbal list-learning task), executive planning (Switching of attention test, Verbal interference test, Maze test, Go-no-go test), and attention (Digit span test, Continuous performance test). A total thinking score will be calculated.
  Z score was calculated, providing a uniform comparison of the raw scores to a normative database, regardless of the original unit of measure used.
  The Z scores have a normative average of 0, with a standard deviation of 1, and no upper of lower limit. Positive values reflect better than average performance, and negative values reflect poorer than average performance.
Time Frame: pre intervention, post 5 weeks intervention, follow-up after 6 months
Measure: Median (Inter-Quartile Range); unit: z-score
Arm/Group | TECH Protocol | Standard Care or Active Standard Care
Number analyzed (Participants) | 30 | 31
z-score
  Pre intervention | -0.6 [-1.1 to -0.3] | -0.9 [-1.2 to -0.5]
  Post 5 weeks intervention | -0.7 [-0.9 to -0.2] | -0.9 [-1.2 to -0.4]
  Follow up after 6 months | -0.7 [-1.1 to -0.3] | -0.7 [-1.2 to -0.4]

3. Secondary Outcome: General Self-Efficacy Scale
Description: Designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life. It consists 10 statements such as 'I can solve most problems if I invest the necessary effort'. Possible responses are scored 1-4 (1 - not at all true to 4 - exactly true), the total score range from 10 to 40. Higher scores represent higher levels of general selfefficacy.
Time Frame: pre intervention, post 5 weeks intervention, follow-up after 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | TECH Protocol | Standard Care or Active Standard Care
Number analyzed (Participants) | 30 | 31
units on a scale
  Pre intervention | 35.0 [30.7 to 37.0] | 35.0 [30.0 to 37.0]
  Post 5 weeks intervention | 34.5 [30.0 to 36.5] | 33.0 [28.0 to 37.0]
  Follow up after 6 months | 35.0 [30.7 to 37.2] | 34.0 [29.0 to 37.0]

4. Secondary Outcome: The 12-Item Short Form Health Survey (SF-12)
Description: SF-12 includes 12 questions from the SF-36 Health Survey. The SF-36 is a widely used and investigated, and validated instrument for measuring quality of life. The SF-12 was developed using normative data for the SF-36 in the United States. The shorter version designed to reproduce the Physical and the Mental Components Summary scores.
  A greater score indicates better health measures. The Physical Composite and Mental Composite will be calculated.
  Scores range from 0 to 100 for each subscale, with higher scores indicating better physical and mental health functioning
Time Frame: pre intervention, post 5 weeks intervention, follow-up after 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | TECH Protocol | Standard Care or Active Standard Care
Number analyzed (Participants) | 30 | 31
units on a scale
  Physical Composite Pre intervention | 29.5 [24.9 to 29.5] | 29.5 [24.9 to 29.5]
  Physical Composite Post 5 weeks intervention | 29.5 [23.8 to 29.5] | 29.5 [24.9 to 29.5]
  Physical Composite Follow up after 6 months | 29.5 [24.9 to 29.5] | 29.5 [24.9 to 29.5]
  Mental Composite Pre intervention | 46.2 [40.1 to 52.3] | 46.2 [46.2 to 52.3]
  Mental Composite Post 5 weeks intervention | 52.3 [44.7 to 52.3] | 46.2 [46.2 to 52.3]
  Mental Composite Follow up after 6 months | 52.3 [40.1 to 52.3] | 46.2 [46.2 to 46.2]

5. Other Pre Specified Outcome: The Geriatric Depression Scale (GDS)
Description: Valid and reliable self-rating screening tool developed to detect depressive symptoms in elderly (D'ath, Katona, Mullan, Evans, & Katona, 1994; Lesher & Berryhill, 1994). The questionnaire includes 15 yes/no statements and takes up to10 minutes to complete.
  Total score ranges from 0-15. A higher score indicates a worse emotional state. Score above 10 points indicates the presence of depressive symptoms (Yesavage et al., 1983).
Time Frame: Pre intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TECH Protocol | Standard Care or Active Standard Care
Number analyzed (Participants) | 30 | 31
units on a scale | 2.8 (1.8) | 2.7 (20.)

6. Other Pre Specified Outcome: Structural and Functional Magnetic Resonance Imaging (MRI)
Description: Changes in brain volume, activity, and white-matter integrity will be assessed by MRI whole brain scanning. MRI scans will be performed on a 3T Prisma Siemens scanner at the Alfredo Federico Strauss Center for Computational Neuroimaging at Tel Aviv University. The MRI scans will include: two short structural assessments - magnetization prepared - rapid gradient echo (MP-RAGE) and fluid-attenuated inversion recovery (FLAIR) - diffusion tensor imaging (DTI) and functional magnetic resonance imaging (f-MRI) (while participants perform the N-back test).
  12 Participants allocated to the TECH intervention (experimental group) will be offered to undergo pre and post MRI scans.
Time Frame: pre, post
Reporting Status: Not Posted

7. Other Pre Specified Outcome: The Tower of Hanoi (ToH) Task - Nomber of Moves
Description: A commonly used goal-directed measure assessing problem-solving, and specifically, planning. A computerized version of the task was used (http://vornlocher.de/tower).The participants completed the first two (out of six) levels of the task. the number of moves per level were recorded. less moves considered better.
Time Frame: pre intervention, post 5 weeks intervention, follow-up after 6 months
Measure: Mean (Standard Deviation); unit: Nomber of moves
Arm/Group | TECH Protocol | Standard Care or Active Standard Care
Number analyzed (Participants) | 30 | 31
Nomber of moves
  level 1 moves pre | 10.3 (3.3) | 14.0 (9.6)
  level 1 moves post | 10.4 (3.6) | 11.1 (6.9)
  level 1 moves follow-up | 9.1 (2.5) | 12.5 (7.9)
  level 2 moves pre | 24.0 (9.2) | 24.1 (7.4)
  level 2 moves post | 24.4 (9.2) | 25.4 (7.8)
  level 2 moves follow up | 24.4 (13.0) | 23.4 (7.1)

8. Other Pre Specified Outcome: The Tower of Hanoi (ToH) Task- Complition Time
Description: A commonly used goal-directed measure assessing problem-solving, and specifically, planning. A computerized version of the task was used (http://vornlocher.de/tower).The participants completed the first two (out of six) levels of the task. the time for completion (seconds) were recorded. Shorter time for completetion considered better.
Time Frame: pre intervention, post 5 weeks intervention, follow-up after 6 months
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | TECH Protocol | Standard Care or Active Standard Care
Number analyzed (Participants) | 30 | 31
Seconds
  level 1 completion time pre | 84.9 (51.2) | 98.0 (66.8)
  level 1 completion time post | 60.0 (31.1) | 70.2 (57.3)
  level 1 completion time follow up | 60.0 (44.9) | 89.7 (67.9)
  level 2 completion time pre | 147.5 (59.5) | 138.3 (55.9)
  level 2 completion time post | 148.9 (78.5) | 132.7 (70.1)
  level 2 completion time follow up | 143.9 (73.2) | 123.0 (63.3)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | TECH Protocol | Standard Care or Active Standard Care
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 0/30 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT02955277/Prot_SAP_000.pdf